CLINICAL TRIAL: NCT02773238
Title: Personalized Radiation Therapy Through Functional Lung Avoidance and Response-Adaptive Dose Escalation: Utilizing Multimodal Molecular Imaging to Improve the Therapeutic Ratio (FLARE RT)
Brief Title: FLARE RT for Patients With Stage IIB-IIIB Non-small Cell Lung Cancer: Personalizing Radiation Therapy Using PET/CT and SPECT/CT Imaging
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jing Zeng, Professor, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9599; NCI-2016-00543 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9599 (Other: Fred Hutch/University of Washington Cancer Consortium); R01CA204301 (NIH); RG3116002 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2016-04-28; First posted 2016-05-16 (Estimated); Results first posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-07

CONDITIONS: Stage IIB Lung Non-Small Cell Carcinoma AJCC v7; Stage IIIA Lung Non-Small Cell Cancer AJCC v7; Stage IIIB Lung Non-Small Cell Cancer AJCC v7
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Fluorodeoxyglucose F18; Magnetic Resonance Spectroscopy; Radiotherapy; Radiation; X-Rays; Photons; Technetium Tc 99m Aggregated Albumin; Technetium Tc 99m Sulfur Colloid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): Patients undergo functional avoidance radiation therapy during weeks 1-3. Patients undergo fludeoxyglucose F-18 FDG PET/CT at baseline, 3 weeks, and 3 months post-radiation therapy and undergo technetium Tc-99m albumin aggregated (99mTc-MAA) and technetium Tc-99m sulfur colloid SPECT/CT radiation therapy at baseline and 3 months post-radiation therapy. Baseline PET/CT must be performed at University of Washington Medical Center/Seattle Cancer Care Alliance and be within one month of treatment start, therefore some patients may need to repeat a baseline PET/CT if their PET/CT is from an outside institution or > 1 month old. Patients not responding to treatment at 3 weeks, will receive an increased daily radiation therapy dosage.
  Interventions: Procedure: Computed Tomography; Radiation: Fludeoxyglucose F-18; Other: Laboratory Biomarker Analysis; Procedure: Positron Emission Tomography; Radiation: Radiation Therapy; Procedure: Single Photon Emission Computed Tomography; Radiation: Technetium Tc-99m Albumin Aggregated; Radiation: Technetium Tc-99m Sulfur Colloid

INTERVENTIONS:
Procedure: Computed Tomography — Undergo FDG PET/CT
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; computerized tomography; CT; CT SCAN; tomography
Procedure: Computed Tomography — Undergo Tc-99m MAA or Tc-99m DTPA
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; computerized tomography; CT; CT SCAN; tomography
Radiation: Fludeoxyglucose F-18 — Undergo FDG PET/CT
  Other Names: 18FDG; FDG; fludeoxyglucose F 18; Fludeoxyglucose F18; Fluorine-18 2-Fluoro-2-deoxy-D-Glucose; Fluorodeoxyglucose F18
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Positron Emission Tomography — Undergo FDG PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging
Radiation: Radiation Therapy — Undergo functional avoidance radiation therapy
  Other Names: Cancer Radiotherapy; Irradiate; Irradiated; irradiation; RADIATION; Radiotherapeutics; radiotherapy; RT; Therapy, Radiation
Procedure: Single Photon Emission Computed Tomography — Undergo Tc-99m MAA or Tc-99m Undergo Tc-99m sulfur colloid SPECT/CT
  Other Names: Medical Imaging, Single Photon Emission Computed Tomography; Single Photon Emission Tomography; single-photon emission computed tomography; SPECT; SPECT imaging; SPECT SCAN; SPET; tomography, emission computed, single photon; Tomography, Emission-Computed, Single-Photon
Radiation: Technetium Tc-99m Albumin Aggregated — Undergo Tc-99m MAA SPECT/CT
  Other Names: Tc 99m-labeled MAA; Technetium Tc 99m-Labeled Macroaggregated Albumin
Radiation: Technetium Tc-99m Sulfur Colloid — Undergo Tc-99m sulfur colloid
  Other Names: Tc 99m sulfur colloid; Tc-99m SC; technetium Tc 99m sulfur colloid

SUMMARY:
This phase II trial studies how well positron emission tomography (PET)/computed tomography (CT) and single positron emission computed tomography (SPECT)/CT imaging works in improving radiation therapy treatment in patients with stage IIB-IIIB non-small cell lung cancer. PET/CT imaging mid-way through treatment may be able to accurately show how well radiation therapy and chemotherapy are working. SPECT/CT imaging may be able to tell which parts of the lung tissue are healthier than others. Based on the result of the imaging, treatment adjustments may be made to the radiation therapy to improve survival and decrease toxicity.

DETAILED DESCRIPTION:
OUTLINE: This is a dose-escalation study of radiation therapy.

Patients undergo functional avoidance radiation therapy during weeks 1-3. Patients undergo fludeoxyglucose F-18 FDG PET/CT at baseline, 3 weeks, and 3 months post-radiation therapy and undergo technetium Tc-99m albumin aggregated (99mTc-MAA) and technetium Tc-99m sulfur colloid SPECT/CT radiation therapy at baseline and 3 months post-radiation therapy. Baseline PET/CT must be performed at University of Washington Medical Center/Seattle Cancer Care Alliance and be within one month of treatment start, therefore some patients may need to repeat a baseline PET/CT if their PET/CT is from an outside institution or > 1 month old. Patients not responding to treatment at 3 weeks, will receive an increased daily radiation therapy dosage.

After completion of study treatment, patients are followed up for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically proven (either histologic or cytologic) diagnosis of stage IIB-IIIB non-small cell lung cancer (NSCLC); according to American Joint Committee on Cancer (AJCC) staging, 7th edition

  * Staging workup must include: brain imaging (CT head or magnetic resonance imaging [MRI] brain) and PET/CT
  * Pleural effusions must have cytology to rule out malignant involvement unless too small to undergo thoracentesis per radiology
* Patients must be considered unresectable or inoperable
* Patient must not have received prior radiation for this lung cancer
* Patients must be having concurrent chemotherapy
* Nodal recurrences can be treated on this protocol but prior curative surgery for lung cancer must have been at least 6 months prior to the nodal recurrence
* Patients must have measurable or evaluable disease that is FDG avid with standardized uptake value (SUV) > 3 on PET/CT
* Zubrod performance status 0-1
* PFTs including forced expiratory volume in 1 second (FEV1) within 26 weeks prior to registration; for FEV1, the best value obtained pre- or post-bronchodilator must be >= 0.8 liters/second or >= 50% predicted
* Blood cell count (CBC)/differential obtained within 8 weeks prior to registration on study
* Absolute neutrophil count (ANC) >= 1,800 cells/mm^3
* Platelets >= 100,000 cells/mm^3
* Hemoglobin >= 10.0 g/dl (Note: The use of transfusion or other intervention to achieve hemoglobin (Hgb) >= 10.0 g/dl is acceptable)
* Serum creatinine within normal institutional limits or creatinine clearance >= 40 ml/min
* Bilirubin must be within or below normal institutional limits
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 2.5 x the institutional upper limit of normal (IULN)
* Patient must sign study specific informed consent prior to study entry

Exclusion Criteria:

* > 10% unintentional weight loss within the past month
* Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 3 years; non-invasive conditions such as carcinoma in situ of the breast, oral cavity, or cervix are all permissible
* Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields
* Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2016-05-20 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jing Zeng, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (2):
- United States (2):
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington
  - SCCA Proton Therapy Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Duan C, Liu Q, Wang J, Tong Q, Bai F, Han J, Wang S, Hippe DS, Zeng J, Bowen SR. GWO+RuleFit: rule-based explainable machine-learning combined with heuristics to predict mid-treatment FDG PET response to chemoradiation for locally advanced non-small cell lung cancer. Phys Med Biol. 2024 Jul 23;69(15):10.1088/1361-6560/ad6118. doi: 10.1088/1361-6560/ad6118. PMID 38981590
- [Derived] Horn KP, Thomas HMT, Vesselle HJ, Kinahan PE, Miyaoka RS, Rengan R, Zeng J, Bowen SR. Reliability of Quantitative 18F-FDG PET/CT Imaging Biomarkers for Classifying Early Response to Chemoradiotherapy in Patients With Locally Advanced Non-Small Cell Lung Cancer. Clin Nucl Med. 2021 Nov 1;46(11):861-871. doi: 10.1097/RLU.0000000000003774. PMID 34172602
- [Derived] Duan C, Chaovalitwongse WA, Bai F, Hippe DS, Wang S, Thammasorn P, Pierce LA, Liu X, You J, Miyaoka RS, Vesselle HJ, Kinahan PE, Rengan R, Zeng J, Bowen SR. Sensitivity analysis of FDG PET tumor voxel cluster radiomics and dosimetry for predicting mid-chemoradiation regional response of locally advanced lung cancer. Phys Med Biol. 2020 Oct 7;65(20):205007. doi: 10.1088/1361-6560/abb0c7. PMID 33027064
- [Derived] Bowen SR, Hippe DS, Chaovalitwongse WA, Duan C, Thammasorn P, Liu X, Miyaoka RS, Vesselle HJ, Kinahan PE, Rengan R, Zeng J. Voxel Forecast for Precision Oncology: Predicting Spatially Variant and Multiscale Cancer Therapy Response on Longitudinal Quantitative Molecular Imaging. Clin Cancer Res. 2019 Aug 15;25(16):5027-5037. doi: 10.1158/1078-0432.CCR-18-3908. Epub 2019 May 29. PMID 31142507

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment
Started | 51
Completed | 47
Not Completed | 4
Not completed — Lack of Efficacy | 4

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.2 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 36
  More than one race | 0
  Unknown or Not Reported | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 51

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS) Rate
Description: Final statistical analyses of OS will consist of Kaplan-Meier estimation.
Time Frame: At 2 years
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Treatment
Number analyzed (Participants) | 51
percentage of patients | 54.2 [41.8 to 70.4]

2. Secondary Outcome: Radiation Pneumonitis Defined as Common Terminology Criteria for Adverse Events Version 4 Grade 2 or Higher Pneumonitis
Description: Common Terminology Criteria for Adverse Events version 4, grade 2 or higher pneumonitis is defined as breathing problems after radiation treatment requiring medications for treatment (grade 2), oxygen use (grade 3), hospitalization (grade 4), or leading to death (grade 5). Clinical studies commonly report how many patients that develop pneumonitis as a result of radiation treatment, which is usually within the first 3 months after radiation.
Time Frame: Up to 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 51
Participants | 17

3. Secondary Outcome: Local-Regional Progression as Defined by Response Evaluation Criteria In Solid Tumors (RECIST) Criteria
Description: Intrathoracic progression of lung tumors assessed by post-radiotherapy computed tomography. Progression will be defined by RECIST criteria. Final statistical analyses of local-regional progression cumulative incidence will consist of Fine-Gray estimation with death and distant metastasis as competing risks.
Time Frame: At 1 year
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Treatment
Number analyzed (Participants) | 51
percentage of patients | 12.2 [4.9 to 23.2]

4. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival will be assessed by post-radiotherapy computed tomography. Progression will be defined by RECIST criteria. Final statistical analyses of PFS will consist of Kaplan-Meier estimation.
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Treatment
Number analyzed (Participants) | 51
percentage of patients | 53.1 [40.9 to 69]

5. Secondary Outcome: Change in Pulmonary Function-forced Expiratory Volume in 1 Second (FEV1)
Description: Pulmonary function tests (FEV1, liters) will be performed and change over time will be evaluated.
Time Frame: Baseline to 3 months post-radiation therapy
Population: 51 patient had pre-radiation PFTs done, but only 45 patients had 3-months post-radiation PFTs performed. Patients either withdrew from study due to cancer progression or declined the repeat testing.
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Treatment
Number analyzed (Participants) | 45
liters | -0.15 (0.09)

6. Secondary Outcome: Change in Pulmonary Function (Diffusing Capacity of the Lungs for Carbon Monoxide [DLCO])
Description: Pulmonary function tests (DLCO, % predicted) will be performed and change over time will be evaluated.
Time Frame: Baseline to 3 months post-radiation therapy
Population: Only 45 patients went through both baseline and 3-months post-radiation testing.
Measure: Mean (Standard Deviation); unit: percentage of predicted lung function
Arm/Group | Treatment
Number analyzed (Participants) | 45
percentage of predicted lung function | -8 (5.2)

ADVERSE EVENTS:
Time Frame: Adverse events were collected during radiation treatment weekly during physician visits, and then monthly after radiation treatment was completed for 3 months.
Description: CTCAE v4 was used to grade adverse events for up to 3 months after completion of radiation. Survival was monitored for up to 2 years after end of radiation.
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 24/51
Serious Adverse Events (participants affected / at risk) | 6/51
Other Adverse Events (participants affected / at risk) | 49/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=51)
Pneumonitis Grade 3+ (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Esophagitis Grade 3+ (Gastrointestinal disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=51)
Pneumonitis Grade 2 (Respiratory, thoracic and mediastinal disorders) | 15 (15)
Esophagitis Grade 2 (Gastrointestinal disorders) | 30 (30)
Dermatitis Grade 2 (Skin and subcutaneous tissue disorders) | 5 (5)
Fatigue Grade 2 (General disorders) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-26): https://cdn.clinicaltrials.gov/large-docs/38/NCT02773238/Prot_SAP_000.pdf